CLINICAL TRIAL: NCT01354054
Title: Effects of a Single Treatment of High or Low Frequency TENS on Pain, Hyperalgesia and Function in Patients With Knee Osteoarthritis
Brief Title: TENS Effectiveness and Knee Osteoarthritis in Humans
Acronym: TOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Barbara Rakel, PhD, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TENS/tops/sluka/rakel
Record Dates: First submitted 2011-05-09; First posted 2011-05-16 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Knee Osteoarthritis
Keywords: Knee OA; TENS
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High frrequency TENS (Experimental): 100 Hz TENS, 100 usec
  Interventions: Procedure: High Frequency TENS
- Low frequency TENS (Experimental): 4 Hz, 100 usec TENS
  Interventions: Procedure: Low frequency TENS
- Placebo TENS (Experimental): 100 Hz, 100 usec, set at motor minus 10% then ramps to off in 45 sec, 40 minutes
  Interventions: Procedure: Placebo TENS
- Control (No Intervention): Age matched controls, no intervention

INTERVENTIONS:
Procedure: High Frequency TENS — 100 usec, 100 Hz, pulse amplitude motor - 10%, 30-40 minutes
  Other Names: Electrical stimulation
  Arms: High frrequency TENS
Procedure: Low frequency TENS — 100 usec, 4 Hz, pulse amplitude motor - 10%, 30-40 minutes
  Other Names: Electrical stimulation
  Arms: Low frequency TENS
Procedure: Placebo TENS — 100 usec, 100 Hz, motor - 10%, pulse amplitude adjusted and maintained for 30 seconds then ramping down to zero in 15 seconds
  Other Names: Placebo electrical stimulation
  Arms: Placebo TENS

SUMMARY:
TENS is a non pharmacological intervention to control pain. Both high (>50 Hz) and low (<10 Hz) frequency TENS are used in the clinic and it is thought that each type works through different mechanisms (see for review Sluka and Walsh, 2003). Hyperalgesia, an increased response to a noxious stimuli, is one component of pain and occurs both at the site of injury, primary hyperalgesia, and outside the site of injury, secondary hyperalgesia. Recent studies in animals with arthritis of the knee show that low and high frequency TENS differentially modulate primary and secondary hyperalgesia.

Therefore the investigators hypothesize that TENS will reduce hyperalgesia and pain with movement resulting in increased function.

DETAILED DESCRIPTION:
The following specific aims will address this hypothesis:

Specific Aim 1 will compare the effect of high frequency TENS, low frequency TENS, and placebo TENS in patients with osteoarthritis on a variety of outcome measures: primary and secondary hyperalgesia, subjective pain scores, and function.

Specific Aim 2 will determine the relationships among these multiple pain measures in people with osteoarthritis, and compare to age matched controls.

Specific Aim 3 will determine the genetic variability as it relates to osteoarthritis pain and response to TENS treatment

Specific Aim 4 will determine how body composition (BMI, fat mass, percent fat, lean mass, and bone mass) impacts the effectiveness of TENS

One of the long-term goals of the investigators is to determine the clinical effectiveness of non-pharmacological treatments for pain, like TENS. These studies will begin to address this issue by examining effects of TENS on a variety of outcome measures in patients with a specific controlled condition (i.e., knee osteoarthritis). This research is innovative because it will be the first to systematically examine the effects of TENS on a variety of physiological parameters (primary and secondary hyperalgesia) and clinical outcome measures (resting pain, movement-evoked pain, function) in a common, painful and limiting condition that is frequently seen in physical therapy clinics. These studies will further allow us to translate basic science experiments previously performed in animal models of arthritis to the clinic. This information is expected to assist the clinician in the treatment choice for a particular patient and guide future clinical research.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of medial compartment knee osteoarthritis
* 18 and 60 years of age
* being able to ambulate to the mail box and back
* stable medication schedule over the last three weeks
* pain rating > 3 on a 0-10 scale when verbally asked to rate knee pain in the weight bearing position
* normal L1-S2 dermatomal screen and normal great toe and thumb proprioception.

Exclusion Criteria:

* Knee surgery in the last six months
* Knee injection in the last four weeks
* serious medical condition, uncontrolled diabetes mellitus, hypertension
* dementia or cognitive impairment
* permanent lower extremity sensory
* prior TENS use

Ages: 30 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold | 3 hours
  A handheld digital pressure algometer (Somedic AB, Farsta, Sweden), was used to assess PPT with the 1 cm2 circular probe. Pressure was applied at 40 kPa/s and patients were instructed to press the hand held response switch when the sensation first became painful. Familiarization with the proceedure was accomplished with testing on the non-dominant forearm of each subject. Following this familiarization procedure, PPTs were assessed at the knee and anterior tibialis muscle bilaterally. An average of the three trials at each test site was used for analysis.
Timed Up and Go test | 3 hours
  The TUG is a standardized test where on command subjects arise from a chair with no arm rest, ambulate 9.8 feet as quickly and safely as possible, turn, ambulate back, turn and return to sitting in the chair. The walking distance was measured in advance and marked on the floor with tape marks well visualized by subjects. Subjects were timed in a standardized fashion from the moment the upper back left the chair until return to full sitting position with back in contact with the chair.
Pain Intensity measures | 3 hours
  Subjects were asked to rate their pain intensity on a horizontal 100 mm Visual Analog Scale (VAS). The anchors utilized were "no pain" and "worst imaginable pain". VAS measures were taken at rest, during the TUG, during the HTS, and cutaneous mechanical pain testing.
Thermal Pain threshold (HPT) and Temporal summation (HTS) | 3 hours
  The TSA II NeuroSensory Analyzer was used to assess (HPT)and (HTS). For both measures, the 5 cm2 probe was placed and initial temperature was set at 37oC, and increased at 1 °C/s to a maximum of 52 oC. Subjects indicated when they first felt pain by using the remote patient switch which recorded the temperature . For temporal summation (HTS), a tonic heat stimulus of 45.5 oC was applied for 20 s. After building to the 45.5 oC in the first 5 s, subjects rated pain caused by this stimulus on a 10 cm visual analog scale every 5s for 15s.
Cutaneous Mechanical Pain testing | 3 hours
  Cutaneous mechanical pain thresholds were assessed with a series of von Frey filaments (North Coast Medical, Gilroy, CA) applied in ascending order from 0.008 to 300 g (0.008, 0.02, 0.04, 0.07, 0.16, 0.4, 0.6, 1.0, 1.4, 2, 4, 6, 8, 10, 15, 26, 60, 100, 180, 300 g). In addition, the subjects rated their pain on a 100 mm VAS in response to application of a 6 g von Frey filament at the six sites bilaterally.

CONTACTS AND LOCATIONS:
Overall Officials: Barbarb A Rakel, PhD, Principal Investigator — University of Iowa College of Nursing; Kathleen A Sluka, PhD, Principal Investigator — University of Iowa Physical Therapy and Rehabilitation Science Graduate Program
Locations (3):
- University of Iowa, Iowa City, Iowa, United States
- Department of Physical Therapy Federal university of Sergipe, Aracaju, Brazil
- Health and Rehabilitation Science Research Institute, University of Ulster , UK, Newtownabbey, Northern Ireland, United Kingdom

REFERENCES:
- [Background] Sluka KA, Walsh D. Transcutaneous electrical nerve stimulation: basic science mechanisms and clinical effectiveness. J Pain. 2003 Apr;4(3):109-21. doi: 10.1054/jpai.2003.434. PMID 14622708
- [Derived] Vance CG, Rakel BA, Blodgett NP, DeSantana JM, Amendola A, Zimmerman MB, Walsh DM, Sluka KA. Effects of transcutaneous electrical nerve stimulation on pain, pain sensitivity, and function in people with knee osteoarthritis: a randomized controlled trial. Phys Ther. 2012 Jul;92(7):898-910. doi: 10.2522/ptj.20110183. Epub 2012 Mar 30. PMID 22466027